CLINICAL TRIAL: NCT00226343
Title: Phase 4 Study: Double-blind Placebo-controlled Trial of Depakote-ER for Depressive and Anxiety Symptoms in Non-refractory Bipolar Depression
Brief Title: Depakote-ER for Depressive and Bipolar Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHA-IRB-0007/07/03
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Valproic Acid

STUDY DESIGN:
Oversight: FDA-regulated Device: No

INTERVENTIONS:
Drug: Depakote-ER

SUMMARY:
Obtain information using a randomized treatment to assess the antidepressant and anxiolytic efficacy of divalproex vs. placebo for nonrefractory bipolar patients with major depressive episodes.

DETAILED DESCRIPTION:
Study is 6 weeks long, with 7 clinical visits.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of bipolar disorder type I or II, non refractory, non-psychotic; females must be nonpregnant/nonlactating; sexually active females must use adequate contraception; MRS < 12; MADRS > 17; no other baseline mood stabilizing drugs, antidepressants or antipsychotics

Exclusion Criteria:

* Active substance abuse or dependence in the past month; medically unstable condition; previously intolerance to valproate; past hepatitis B or C, or serious liver disease; serious suicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-08; Primary Completion 2006-01 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Anxiety and Depressive Symptom severity

CONTACTS AND LOCATIONS:
Overall Officials: Robert T Dunn, MD, PhD, Principal Investigator — Cambridge Health Alliance

REFERENCES:
- [Derived] Ghaemi SN, Gilmer WS, Goldberg JF, Zablotsky B, Kemp DE, Kelley ME, Bauer AD, Fleck J, Filkowski MM, Stan VA, Dunn RT. Divalproex in the treatment of acute bipolar depression: a preliminary double-blind, randomized, placebo-controlled pilot study. J Clin Psychiatry. 2007 Dec;68(12):1840-4. doi: 10.4088/jcp.v68n1203. PMID 18162014